CLINICAL TRIAL: NCT05718687
Title: A PHASE 1 STUDY TO ASSESS THE MASS BALANCE, EXCRETION, AND PHARMACOKINETICS OF [14C]-GBT021601, AN ORAL HEMOGLOBIN SPOLYMERIZATION INHIBITOR, IN HEALTHY PARTICIPANTS
Brief Title: A GBT021601 ADME Microtracer Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GBT021601-013; C5351003 (Other: Alias Study Number); 2022-003108-34 (EudraCT Number)
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): open-label GBT021601
  Interventions: Drug: GBT021601

INTERVENTIONS:
Drug: GBT021601 — Single oral dose of 200 mg GBT021601, containing ~74 kBq (~2 µCi) of [14C]-GBT021601

SUMMARY:
An Open-label Study of GBT021601 in 8 to 10 healthy male or female participants to evaluate the absorption, distribution, metabolism, and excretion (ADME) of GBT021601.

DETAILED DESCRIPTION:
This is an open-label Study administering GBT021601 as a single oral dose of 200 mg in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): 18.0 to 27.0 kg/m2, inclusive, at screening.
* Body weight ≥ 50 kg at screening
* Females must be nonlactating and nonpregnant (as confirmed by a negative serum pregnancy test at screening and admission for all females), or of nonchildbearing potential (ie, either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1 year postmenopausal [defined as at least 12 months no menses, and confirmed by a follicle-stimulating hormone test, at screening]).
* Creatinine clearance (glomerular filtration rate) as estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula: ≥90 mL/min, at screening.

Exclusion Criteria:

* History or presence of conditions which, in the opinion of the Investigator, are known to interfere with the ADME of drugs, such as previous surgery on the gastrointestinal tract (including removal of parts of the stomach, bowel, liver, gall bladder, or pancreas). Participants who have a history of appendectomy are eligible for enrollment.
* History of chronic constipation, or recent complaints of an irregular defecation
* Significant and/or acute illness at screening or within 5 days prior to study drug administration that may impact safety assessments, in the opinion of the Investigator.
* Known personal or family history of congenital long QT syndrome or known family history of sudden death.
* Participation in another ADME study with a radiation burden >0.1 mSv in the period of 1 year prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- ICON Early Phase Clinic, LLC, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT021601-013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 participants were enrolled in this study.
Groups:
- GBT021601+[14C]-GBT021601: Participants were administered a single 200 milligrams (mg) oral dose of GBT021601 containing approximately 74 kilobecquerel (kBq) (approximately 2 microcurie [mcCi]) of [14C] labelled GBT021601 on Day 1.
Period: Overall Study
Arm/Group | GBT021601+[14C]-GBT021601
Started | 9
Completed | 6
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had received 1 dose of GBT021601.
Groups:
- GBT021601+[14C]-GBT021601: Participants were administered a single 200 mg oral dose of GBT021601 containing approximately 74 kBq (approximately 2 mcCi) of [14C] labelled GBT021601 on Day 1.
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.6 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at Predose
Time Frame: Predose (within 60 minutes prior to GBT021601 dosing)
Population: Pharmacokinetic (PK) analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity in whole blood or plasma.
Measure: Mean (Standard Deviation); unit: Microgram/ milliliter (mcg/mL)
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Microgram/ milliliter (mcg/mL)
  Whole blood | NA (NA) — Mean and SD were not estimated as data was below the lower limit of quantification (LLOQ),
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.

2. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at Predose
Description: Data reported in microgram equivalent per milliliter (mcgEq/mL).
Time Frame: Predose (within 60 minutes prior to 14C-GBT021601 dosing)
Population: PK analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity in whole blood or plasma.
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole blood | 0 (0)
  Plasma | 0 (0)

3. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 0.25 Hours
Time Frame: 0.25 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole blood | 6.368 (5.4178)
  Plasma | 0.46267 (0.373675)

4. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentrations in Whole Blood and Plasma at 0.25 Hours
Time Frame: 0.25 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 5.8206 (4.64396)
  Plasma | 0.84819 (0.595349)

5. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 0.50 Hours
Time Frame: 0.50 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 17.33 (4.122)
  Plasma | 1.2338 (0.37097)

6. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 0.50 Hours
Time Frame: 0.50 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 16.45 (4.348)
  Plasma | 2.345 (0.6467)

7. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 1 Hours
Time Frame: 1 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 29.37 (4.520)
  Plasma | 1.433 (0.1997)

8. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 1 Hours
Time Frame: 1 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 27.24 (4.590)
  Plasma | 2.913 (0.4117)

9. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 2 Hours
Time Frame: 2 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 31.92 (6.544)
  Plasma | 0.9228 (0.21798)

10. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 2 Hours
Time Frame: 2 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 29.52 (5.586)
  Plasma | 2.089 (0.4195)

11. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 3 Hours
Time Frame: 3 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 31.92 (6.544)
  Plasma | 0.5974 (0.13629)

12. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 3 Hours
Time Frame: 3 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 29.78 (5.540)
  Plasma | 1.502 (0.2753)

13. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 4 Hours
Time Frame: 4 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 34.96 (6.738)
  Plasma | 0.4539 (0.14820)

14. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 4 Hours
Time Frame: 4 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 31.23 (6.483)
  Plasma | 1.2243 (0.32688)

15. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 6 Hours
Time Frame: 6 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 34.84 (7.996)
  Plasma | 0.3013 (0.07405)

16. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 6 Hours
Time Frame: 6 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 31.51 (7.104)
  Plasma | 0.8534 (0.19276)

17. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 8 Hours
Time Frame: 8 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 36.00 (8.979)
  Plasma | 0.2267 (0.06210)

18. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 8 Hours
Time Frame: 8 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 31.53 (8.016)
  Plasma | 0.6592 (0.13795)

19. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 12 Hours
Time Frame: 12 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 36.49 (10.844)
  Plasma | 0.1986 (0.05917)

20. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 12 Hours
Time Frame: 12 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 32.95 (7.459)
  Plasma | 0.5064 (0.11455)

21. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 24 Hours
Time Frame: 24 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 37.53 (8.855)
  Plasma | 0.1479 (0.03685)

22. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 24 Hours
Time Frame: 24 hours post dosing on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 33.62 (7.819)
  Plasma | 0.3256 (0.06395)

23. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 48 Hours
Time Frame: 48 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 37.39 (9.904)
  Plasma | 0.1402 (0.02718)

24. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 48 Hours
Time Frame: 48 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 33.29 (7.384)
  Plasma | 0.2207 (0.03853)

25. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 72 Hours
Time Frame: 72 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 35.41 (7.642)
  Plasma | 0.1377 (0.03011)

26. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 72 Hours
Time Frame: 72 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 31.38 (6.475)
  Plasma | 0.1861 (0.03361)

27. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 96 Hours
Time Frame: 96 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 34.67 (7.339)
  Plasma | 0.12923 (0.026617)

28. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 96 Hours
Time Frame: 96 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 30.62 (5.839)
  Plasma | 0.1670 (0.03204)

29. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 144 Hours
Time Frame: 144 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 32.48 (7.257)
  Plasma | 0.11038 (0.016657)

30. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 144 Hours
Time Frame: 144 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 28.81 (5.988)
  Plasma | 0.1434 (0.02345)

31. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 168 Hours
Time Frame: 168 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 32.91 (7.603)
  Plasma | 0.12189 (0.020679)

32. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 168 Hours
Time Frame: 168 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 27.33 (5.329)
  Plasma | 0.1471 (0.03267)

33. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 312 Hours
Time Frame: 312 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 26.59 (5.353)
  Plasma | 0.11109 (0.024207)

34. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 312 Hours
Time Frame: 312 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 23.44 (3.976)
  Plasma | 0.1274 (0.01847)

35. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 480 Hours
Time Frame: 480 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 22.38 (3.991)
  Plasma | 0.08271 (0.014586)

36. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 480 Hours
Time Frame: 480 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 19.30 (2.743)
  Plasma | 0.09706 (0.010952)

37. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 648 Hours
Time Frame: 648 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 18.71 (3.597)
  Plasma | 0.07343 (0.011345)

38. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 648 Hours
Time Frame: 648 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 16.32 (2.161)
  Plasma | 0.08224 (0.007987)

39. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 816 Hours
Time Frame: 816 hours post dosing
Population: PK analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity in whole blood or plasma. Here "Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
mcg/mL
  Whole Blood | 15.20 (1.553)
  Plasma | 0.06894 (0.011486)

40. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 816 Hours
Time Frame: 816 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
mcgEq/mL
  Whole Blood | 12.93 (1.403)
  Plasma | 0.08084 (0.005649)

41. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 984 Hours
Time Frame: 984 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 12.60 (1.715)
  Plasma | 0.05919 (0.006786)

42. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 984 Hours
Time Frame: 984 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 11.087 (1.4815)
  Plasma | 0.06646 (0.005689)

43. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 1320 Hours
Time Frame: 1320 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole Blood | 8.772 (1.1434)
  Plasma | 0.03829 (0.003602)

44. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 1320 Hours
Time Frame: 1320 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole Blood | 7.599 (1.1109)
  Plasma | 0.04387 (0.004128)

45. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 1656 Hours
Time Frame: 1656 hours post dosing
Population: PK analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity in whole blood or plasma. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
mcg/mL
  Whole Blood | 6.253 (0.9576)
  Plasma | 0.02809 (0.005965)

46. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 1656 Hours
Time Frame: 1656 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
mcgEq/mL
  Whole Blood | 5.528 (1.0078)
  Plasma | 0.02835 (0.004387)

47. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 1992 Hours
Time Frame: 1992 hours post dosing
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
mcg/mL
  Whole Blood | 4.283 (0.7310)
  Plasma | 0.01881 (0.003921)

48. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 1992 Hours
Time Frame: 1992 hours post dosing
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
mcgEq/mL
  Whole Blood | 3.667 (0.5431)
  Plasma | 0.01909 (0.004378)

49. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 2328 Hours
Time Frame: 2328 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 6
mcg/mL
  Whole Blood | 2.997 (0.6994)
  Plasma | 0.01407 (0.007193)

50. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 2328 Hours
Time Frame: 2328 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 6
mcgEq/mL
  Whole Blood | 2.677 (0.5212)
  Plasma | 0.013250 (0.0042927)

51. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 2664 Hours
Time Frame: 2664 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 5
mcg/mL
  Whole Blood | 2.290 (0.4786)
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the lower limit of quantification.

52. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 2664 Hours
Time Frame: 2664 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 5
mcgEq/mL
  Whole Blood | 2.064 (0.3699)
  Plasma | 0.008206 (0.0031073)

53. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 3240 Hours
Time Frame: 3240 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 3
mcg/mL
  Whole Blood | 1.1523 (0.38725)
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the lower limit of quantification.

54. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 3240 Hours
Time Frame: 3240 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 3
mcgEq/mL
  Whole Blood | 0.9463 (0.30792)
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.

55. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 3576 Hours
Time Frame: 3576 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 3
mcg/mL
  Whole Blood | 0.6097 (0.52801)
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.

56. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 3576 Hours
Time Frame: 3576 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 3
mcgEq/mL
  Whole Blood | 0.6733 (0.24908)
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.

57. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 4248 Hours
Time Frame: 4248 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 2
mcg/mL
  Whole Blood | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.

58. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 4248 Hours
Time Frame: 4248 hours post dosing
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 2
mcgEq/mL
  Whole Blood | 0.2745 (0.14637)
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.

59. Primary Outcome: GBT021601 Concentration in Whole Blood and Plasma at 4920 Hours
Time Frame: 4920 hours post dosing
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 1
mcg/mL
  Whole Blood | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.

60. Primary Outcome: 14C-GBT021601 Total Radioactivity Concentration in Whole Blood and Plasma at 4920 Hours
Time Frame: 4920 hours post dosing
Population: PK analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity in whole blood or plasma. Here " Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 1
mcgEq/mL
  Whole Blood | 0.2330 (NA) — SD was not estimable as only 1 participant was analyzed.
  Plasma | NA (NA) — Mean and SD were not estimated as data was below the LLOQ.

61. Primary Outcome: Cumulative Amount of [14C]-GBT021601 Total Radioactivity Excreted in Urine and Feces
Description: Data are reported as aggregate of all scheduled time points.
Time Frame: Day 1 (prior to dosing), after dosing from 0-6 hours, 6-12 hrs, 12-24 hrs postdose for urine, 24-hr intervals up to Day 29; 816 hrs , 984 hrs, 1320 hrs, 1656 hrs, 1992 hrs, 2328 hrs, 2664 hrs, 3240 hrs, 3576 hrs, 4248 hrs, and 4920 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram equivalents (mgEq)
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
milligram equivalents (mgEq)
  Urine | 95.23 (10.153)
  Feces | 81.38 (12.668)

62. Primary Outcome: Cumulative Fraction of [14C]-GBT021601 Total Radioactivity Excreted in Urine and Feces
Description: Data are reported as aggregate of all scheduled time points.
Time Frame: as for outcome 61
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of administered drug
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Percentage of administered drug
  Urine | 47.24 (5.036)
  Feces | 40.37 (6.284)

63. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero (0) to 24 Hours (AUC0-24) of GBT021601 in Whole Blood and Plasma
Description: Area under the plasma concentration-time curve up to 24 hours post dose. Data reported in Hour*microgram/millimeter (h*mcg/mL).
Time Frame: Day 1 (prior to dosing) at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
h*mcg/mL
  Whole Blood | 824.1 (22.3)
  Plasma | 7.393 (20.0)

64. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero (0) to 24 Hours (AUC0-24) of 14C-GBT021601 in Whole Blood and Plasma
Description: Area under the plasma concentration-time curve up to 24 hours postdose. Data reported in hour*microgram equivalent/milliliter (h*mcgEq/mL).
Time Frame: Day 1 (prior to dosing) at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
h*mcgEq/mL
  Whole Blood | 741.8 (21.3)
  Plasma | 17.92 (19.2)

65. Primary Outcome: Area Under the Concentration-Time From Time Zero to the Last Measurable Concentration (AUC0-last) of GBT021601 in Whole Blood and Plasma
Time Frame: Day 1 (prior to dosing), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144,168, 312, 480, 648, 816, 984,1320,1656,1992, 2328, 2664, 3240, 3576, 4248 and 4920 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
h*mcg/mL
  Whole blood | 31481.7 (20.9)
  Plasma | 130.35 (16.7)

66. Primary Outcome: Area Under the Concentration-Time From Time Zero to the Last Measurable Concentration (AUC0-last) of 14C-GBT021601 in Whole Blood and Plasma
Time Frame: as for outcome 65
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
h*mcgEq/mL
  Whole blood | 27609.6 (18.5)
  Plasma | 165.7 (13.1)

67. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of GBT021601 in Whole Blood and Plasma
Description: Area under the plasma concentration-time curve from time 0 to infinity calculated as: AUC0-inf=AUC0-t+Clast/kel, where Clast is the last measurable plasma concentration.
Time Frame: as for outcome 65
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
h*mcg/mL
  Whole blood | 35290.5 (12.1)
  Plasma | 150.7 (10.8)

68. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of 14C-GBT021601 in Whole Blood and Plasma
Description: Area under the plasma concentration-time curve from time 0 to infinity calculated as: AUC0-inf=AUC0-t+Clast/kel, where Clast is the last measurable plasma concentration and Kel is apparent terminal elimination rate constant.
Time Frame: as for outcome 65
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
h*mcgEq/mL
  Whole blood | 30636.1 (10.5)
  Plasma | 179.1 (8.8)

69. Primary Outcome: Maximum Observed Concentration (Cmax) of GBT021601 in Whole Blood and Plasma
Time Frame: as for outcome 65
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcg/mL
  Whole blood | 40.06 (27.1)
  Plasma | 1.468 (14.0)

70. Primary Outcome: Maximum Observed Concentration (Cmax) of 14C-GBT021601 in Whole Blood and Plasma
Time Frame: as for outcome 65
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcgEq/mL
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mcgEq/mL
  Whole blood | 34.05 (20.8)
  Plasma | 2.950 (12.5)

71. Primary Outcome: Time to Attain Maximum Observed Concentration (Tmax) of GBT021601 in Whole Blood and Plasma
Time Frame: as for outcome 65
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Hour (h)
  Whole blood | 24.000 [8.00 to 72.03]
  Plasma | 1.000 [0.50 to 1.00]

72. Primary Outcome: Time to Attain Maximum Observed Concentration (Tmax) of 14C-GBT021601 in Whole Blood and Plasma
Time Frame: as for outcome 65
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Hour
  Whole blood | 24.000 [4.00 to 48.00]
  Plasma | 1.000 [0.50 to 1.00]

73. Primary Outcome: Apparent Terminal Elimination Half-Life (t1/2) of GBT021601 in Whole Blood and Plasma
Description: Apparent terminal elimination half-life, calculated as 0.693/kel where kel is Apparent terminal elimination rate constant.
Time Frame: as for outcome 65
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Hour
  Whole blood | 647.8 (84.51)
  Plasma | 707.1 (112.32)

74. Primary Outcome: Apparent Terminal Elimination Half-Life (t1/2) of 14C-GBT021601 in Whole Blood and Plasma
Description: as for outcome 73
Time Frame: as for outcome 65
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Hour
  Whole blood | 654.7 (92.46)
  Plasma | 588.9 (109.92)

75. Primary Outcome: Renal Clearance (CLR) of GBT021601 and 14C-GBT021601 in Urine
Description: Renal clearance was calculated as CLR = Ae0-inf/AUC0-inf. Where Ae indicates Cumulative amount of drug excreted and AUC0-inf indicates Area under the plasma concentration-time curve from time 0 to infinity.
Time Frame: as for outcome 65
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
Liter/hour (L/h) | 0.2755 (12.6)

76. Primary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/F) of GBT021601 in Whole Blood and Plasma
Description: Apparent volume of distribution at terminal phase, calculated as: (CL/F) Apparent total clearance, calculated as dose/AUC0-inf/Kel.
Time Frame: as for outcome 65
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
Liter (L)
  Whole blood | 5.175 (18.3)
  Plasma | 1300.6 (15.5)

77. Primary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/F) of 14C-GBT021601 in Whole Blood and Plasma
Description: as for outcome 76
Time Frame: as for outcome 65
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
Liter
  Whole blood | 5.972 (15.9)
  Plasma | 906.1 (14.4)

78. Primary Outcome: Apparent Total Clearance (CL/F) of GBT021601 in Whole Blood and Plasma
Description: Apparent total clearance, calculated as dose/AUC0-inf.
Time Frame: as for outcome 65
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
L/h
  Whole blood | 0.005713 (12.1)
  Plasma | 1.338 (10.8)

79. Primary Outcome: Apparent Total Clearance (CL/F) of 14C-GBT021601 in Whole Blood and Plasma
Description: Apparent total clearance, calculated as dose/AUC0-inf.
Time Frame: as for outcome 65
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
L/h
  Whole blood | 0.006580 (10.5)
  Plasma | 1.1258 (8.8)

80. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 0-6 Hours
Time Frame: 0-6 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 13.123 (4.5812)
  Feces: number analyzed (Participants) | 0

81. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 6-12 Hours
Time Frame: 6-12 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 16.611 (4.2333)
  Feces: number analyzed (Participants) | 0

82. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 12-24 Hours
Time Frame: 12-24 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 19.70 (4.021)
  Feces: number analyzed (Participants) | 0

83. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 0-24 Hours
Time Frame: 0-24 hours post dose
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 7
mgEq
  Urine: number analyzed (Participants) | 0
  Feces | 0.060486 (0.1389173)

84. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 24 Hours
Time Frame: 24 hours post dose
Population: PK analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity in whole blood or plasma. Here "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 23.19 (4.305)
  Feces: number analyzed (Participants) | 8
  Feces | 24.25 (9.726)

85. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 48 Hours
Time Frame: 48 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 25.50 (4.727)
  Feces: number analyzed (Participants) | 8
  Feces | 33.17 (7.021)

86. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 72 Hours
Time Frame: 72 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 27.55 (5.112)
  Feces: number analyzed (Participants) | 6
  Feces | 35.06 (8.909)

87. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 96 Hours
Time Frame: 96 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 29.35 (5.504)
  Feces: number analyzed (Participants) | 8
  Feces | 37.31 (8.103)

88. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 120 Hours
Time Frame: 120 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 30.97 (5.791)
  Feces: number analyzed (Participants) | 8
  Feces | 40.54 (4.600)

89. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 144 Hours
Time Frame: 144 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 32.88 (6.151)
  Feces: number analyzed (Participants) | 7
  Feces | 39.51 (8.832)

90. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 168 Hours
Time Frame: 168 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 34.82 (6.438)
  Feces | 40.87 (7.673)

91. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 192 Hours
Time Frame: 192 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 36.72 (6.695)
  Feces: number analyzed (Participants) | 8
  Feces | 44.39 (5.139)

92. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 216 Hours
Time Frame: 216 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 38.48 (6.926)
  Feces: number analyzed (Participants) | 7
  Feces | 43.09 (9.219)

93. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 240 Hours
Time Frame: 240 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 40.22 (7.197)
  Feces: number analyzed (Participants) | 8
  Feces | 43.54 (8.212)

94. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 264 Hours
Time Frame: 264 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 41.99 (7.402)
  Feces: number analyzed (Participants) | 8
  Feces | 45.31 (8.482)

95. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 288 Hours
Time Frame: 288 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 43.65 (7.589)
  Feces: number analyzed (Participants) | 8
  Feces | 44.72 (7.324)

96. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 312 Hours
Time Frame: 312 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 45.06 (7.759)
  Feces: number analyzed (Participants) | 7
  Feces | 46.29 (9.018)

97. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 336 Hours
Time Frame: 336 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 46.50 (7.899)
  Feces: number analyzed (Participants) | 7
  Feces | 50.24 (5.880)

98. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 360 Hours
Time Frame: 360 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 47.92 (8.085)
  Feces | 48.56 (8.315)

99. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 384 Hours
Time Frame: 384 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 49.41 (8.242)
  Feces: number analyzed (Participants) | 7
  Feces | 52.20 (6.116)

100. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 408 Hours
Time Frame: 408 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 50.87 (8.418)
  Feces: number analyzed (Participants) | 8
  Feces | 49.97 (9.261)

101. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 432 Hours
Time Frame: 432 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 52.24 (8.469)
  Feces: number analyzed (Participants) | 8
  Feces | 50.84 (9.215)

102. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 456 Hours
Time Frame: 456 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 53.59 (8.564)
  Feces: number analyzed (Participants) | 8
  Feces | 53.99 (6.398)

103. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 480 Hours
Time Frame: 480 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 54.81 (8.616)
  Feces: number analyzed (Participants) | 8
  Feces | 52.89 (9.678)

104. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 504 Hours
Time Frame: 504 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 56.00 (8.649)
  Feces: number analyzed (Participants) | 8
  Feces | 53.22 (9.709)

105. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 528 Hours
Time Frame: 528 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 57.15 (8.734)
  Feces: number analyzed (Participants) | 8
  Feces | 56.23 (6.834)

106. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 552 Hours
Time Frame: 552 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 58.19 (8.845)
  Feces: number analyzed (Participants) | 8
  Feces | 55.14 (9.750)

107. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 576 Hours
Time Frame: 576 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 59.25 (9.013)
  Feces: number analyzed (Participants) | 8
  Feces | 55.39 (9.766)

108. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 600 Hours
Time Frame: 600 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 60.20 (9.159)
  Feces: number analyzed (Participants) | 8
  Feces | 58.26 (7.116)

109. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 624 Hours
Time Frame: 624 hours post dose
Population: as for outcome 84
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 61.13 (9.230)
  Feces: number analyzed (Participants) | 8
  Feces | 57.17 (9.867)

110. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 648 Hours
Time Frame: 648 hours post dose
Population: PK analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity in whole blood or plasma. ere "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 62.18 (9.313)
  Feces: number analyzed (Participants) | 6
  Feces | 59.51 (8.648)

111. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 816 Hours
Time Frame: 816 hours post dose
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
mgEq
  Urine | 67.24 (8.848)
  Feces | 62.99 (11.632)

112. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 984 Hours
Time Frame: 984 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 74.37 (9.568)
  Feces | 67.30 (11.537)

113. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 1320 Hours
Time Frame: 1320 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
mgEq
  Urine | 83.07 (9.068)
  Feces | 72.95 (12.135)

114. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 1656 Hours
Time Frame: 1656 hours post dose
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
mgEq
  Urine | 89.48 (9.168)
  Feces | 76.42 (13.642)

115. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 1992 Hours
Time Frame: 1992 hours post dose
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 8
mgEq
  Urine | 93.46 (9.065)
  Feces | 79.01 (14.557)

116. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 2328 Hours
Time Frame: 2328 hours post dose
Population: PK analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity in whole blood or plasma. Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure, where "Number Analyzed" signifies number of participants evaluable for specified row.
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 6
mgEq
  Urine | 92.85 (7.592)
  Feces: number analyzed (Participants) | 5
  Feces | 84.14 (15.744)

117. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 2664 Hours
Time Frame: 2664 hours post dose
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 2
mgEq
  Urine | 100.08 (12.033)
  Feces | 59.86 (0.613)

118. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 3240 Hours
Time Frame: 3240 hours post dose
Population: PK analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity. Here "Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 3
mgEq
  Urine | 98.36 (10.969)
  Feces | 69.27 (13.344)

119. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 3576 Hours
Time Frame: 3576 hours post dose
Population: PK analysis set included all participants who had received 1 dose of GBT021601 and provided at least 1 measurable post dose PK concentration of GBT021601 or total radioactivity in whole blood or plasma. Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 3
mgEq
  Urine | 98.96 (11.161)
  Feces | 69.62 (13.175)

120. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 4248 Hours
Time Frame: 4248 hours post dose
Population: as for outcome 116
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 2
mgEq
  Urine | 93.30 (3.569)
  Feces: number analyzed (Participants) | 1
  Feces | 85.10 (NA) — SD was not estimable as only 1 participant was analyzed.

121. Primary Outcome: Distribution of 14C- GBT021601 Total Radioactivity in Urine and Feces at 4920 Hours
Time Frame: 4920 hours post dose
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mgEq
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 1
mgEq
  Urine | 96.31 (NA) — SD was not estimable as only 1 participant was analyzed.
  Feces | 63.87 (NA) — SD was not estimable as only 1 participant was analyzed.

122. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) was any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. TEAEs were those which occurred (or worsened) after the dose of study drug during the on-treatment period, defined as the period after the dose of study drug and through the minimum of (Study Day 57, study discontinuation).
Time Frame: From Day 1 up to maximum of Day 57
Population: Safety analysis set included all participants who had received 1 dose of GBT021601.
Measure: Count of Participants; unit: Participants
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Participants | 4

123. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values
Description: Blood and urine samples was collected for clinical laboratory assessments. Clinical Laboratory Values included Clinical chemistry: alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bicarbonate, bilirubin (total, direct, and indirect), blood urea nitrogen, calcium, chloride, creatinine, gamma glutamyl transferase, glucose, lactate dehydrogenase, magnesium, phosphorus, potassium, sodium, total protein, and uric acid. Hematology: leukocytes, erythrocytes, hematocrit, Hb, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count (ie, thrombocytes), RBC count, and white blood cell count etc. Urinalysis: determination of pH and specific gravity, and presence of bilirubin, blood, glucose, ketones, nitrite, protein, leukocytes, and urobilinogen etc. Coagulation, Serology, Drug and alcohol screen and Pregnancy test. Clinical significance was judged by investigator.
Time Frame: Day 1 of dosing to Day 207
Population: Safety analysis set included all participants who had received 1 dose of GBT021601.
Measure: Count of Participants; unit: Participants
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Participants | 0

124. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Values
Description: Systolic and diastolic blood pressure and pulse was recorded after the participant had rested for at least 5 minutes in the supine position. Body temperature and respiratory rate was also measured. Clinical significance was judged by investigator.
Time Frame: Day 1 of dosing to Day 207
Population: Safety analysis set included all participants who had received 1 dose of GBT021601.
Measure: Count of Participants; unit: Participants
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Participants | 0

125. Secondary Outcome: Number of Participants With Clinically Significant ECG Values
Description: Standard 12-lead ECGs were performed after the participant had rested quietly for more than 5 minutes in a supine position utilizing an ECG machine that was equipped with computer-based interval measurements. The following measurement was recorded: the heart rate (of <45 or >100 beats per minute (BPM) , PR interval, QT interval, QT interval corrected using Fridericia's formula (QTcF) of >450 msec for males and >470 msec for females, and QRS duration. Any cardiac rhythm other than sinus rhythm that was interpreted by the Investigator was clinically significant.
Time Frame: Day 1
Population: Safety analysis set included all participants who had received 1 dose of GBT021601.
Measure: Count of Participants; unit: Participants
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Participants | 0

126. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Values
Description: Physical Examination test included body weight and height. physical examination was conducted at screening. Clinical significance was judged by investigator.
Time Frame: Screening (-28 Day to -2 Day, day with respect to dosing)
Population: Safety analysis set included all participants who had received 1 dose of GBT021601.
Measure: Count of Participants; unit: Participants
Arm/Group | GBT021601+[14C]-GBT021601
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to maximum of Day 207
Description: Same event may appear as both non-SAE and SAE, but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set was evaluated.
Arm/Group | GBT021601+[14C]-GBT021601
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GBT021601+[14C]-GBT021601 (N=9)
Headache (Nervous system disorders) | 2
Nausea (Gastrointestinal disorders) | 1
COVID-19 (Infections and infestations) | 1
Animal scratch (Injury, poisoning and procedural complications) | 1
Polymenorrhoea (Reproductive system and breast disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Data for metabolite profiling was not reported for [14C]-GBT021601 in whole blood and plasma because it was planned to be collected as part of separate, pooled analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT05718687/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT05718687/SAP_001.pdf